CLINICAL TRIAL: NCT05428969
Title: A Phase I/II Open-Label Study to Assess the Safety, Tolerability and Preliminary Efficacy of the Clever-1 Antibody Bexmarilimab in Combination With Standard of Care Therapy in Patients With Myelodysplastic Syndrome or Chronic Myelomonocytic Leukemia or Acute Myeloid Leukemia
Brief Title: A Study to Assess Safety, Tolerability and Preliminary Efficacy of Bexmarilimab in Combination With Standard of Care in Patients With Hematological Malignancies
Acronym: BEXMAB
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Faron Pharmaceuticals Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: FP2CLI004; 2021-002104-12 (EudraCT Number)
Record Dates: First submitted 2022-06-15; First posted 2022-06-23 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Acute Myeloid Leukemia; Chronic Myelomonocytic Leukemia; Myelodysplastic Syndromes; Relapsed/Refractory AML
Keywords: Macrophages; Immunotherapy; Hematological; CLEVER-1; bexmarilimab; hematological neoplasms; azacitidine; venetoclax; myeloid cells
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Leukemia, Myelomonocytic, Chronic; Myelodysplastic Syndromes; Hematologic Neoplasms | interventions — bexmarilimab; Azacitidine; venetoclax

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Phase 1 - Intermediate/high risk MDS, CMML 10-19%, MDS/CMML failure to HMA, r/r AML (Experimental): Standard of care azacitidine as per label; bexmarilimab 4 dose levels at once every week (Q1W) followed by once every 2 weeks (Q2W); 28-day cycle
  Interventions: Drug: Bexmarilimab; Drug: Azacitidine
- Phase 1 - Newly diagnosed AML patients non-fit for induction therapy (Experimental): Standard of care azacitidine and venetoclax as per label; bexmarilimab 4 dose levels Q1W followed by Q2W; 28-day cycle
  Interventions: Drug: Bexmarilimab; Drug: Azacitidine; Drug: Venetoclax
- Phase 2 - Intermediate/high risk MDS, CMML, MDS/CMML failure to HMA, r/r AML & newly diagnosed AML (Experimental): Standard of care venetoclax and/or azacitidine as per label plus bexmarilmab
  Interventions: Drug: Bexmarilimab; Drug: Azacitidine; Drug: Venetoclax

INTERVENTIONS:
Drug: Bexmarilimab — Intravenous
  Other Names: FP-1305
Drug: Azacitidine — As per label, subcutaneous
Drug: Venetoclax — Oral
  Other Names: Venclyxto®
  Arms: Phase 1 - Newly diagnosed AML patients non-fit for induction therapy; Phase 2 - Intermediate/high risk MDS, CMML, MDS/CMML failure to HMA, r/r AML & newly diagnosed AML

SUMMARY:
This is a study to assess the safety of increasing dose levels of bexmarilimab when combined with standard of care (SoC) in patients with myelodysplastic syndrome (MDS) or chronic myelomonocytic leukemia (CMML) or acute myeloid leukemia (AML); Phase 1 aims to identify the recommended phase 2 dose (RP2D) of bexmarilimab based on safety, tolerability and pharmacological activity; Phase 2 will investigate the preliminary efficacy of the combination treatment in selected indications from Phase 1.

DETAILED DESCRIPTION:
This is a multicenter Phase 1/2 open-label, study to assess the safety, tolerability and preliminary efficacy of increasing doses of bexmarilimab (FP-1305) in patients with intermediate, high or very high-risk MDS, CMML with 10-19 % marrow blasts, CMML/MDS with failure to hypomethylating agent (HMA), or in patients with newly diagnosed AML non-fit for induction therapy or relapsed/refractory AML. The Phase 1 part of the study will identify a safe and tolerable bexmarilimab dose amongst four predefined dose levels using a bayesian optimal interval (BOIN) dose escalation design to identify the maximum tolerated dose (MTD) of bexmarilimab when administered in combination with SoC.

The Phase 2 of the study is an expansion phase to further evaluate the safety and preliminary efficacy of bexmarilimab treatment at RP2D combined with SoC and will follow a Simon's 2-stage design for each of the indications selected to continue forward from Phase 1. This design allows for the investigation of bexmarilimab activity and preliminary response assessments tailored to each indication and allows early stopping in case of futility using a minimum number of patients. Patients from Phase 1, with the selected indication to be investigated in Phase 2, that have been treated at RP2D may be counted towards the number of patients for Phase 2.

Both study phases consist of a screening period, a treatment period, an end of treatment (EoT) as safety follow-up and disease progression/survival follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Patient ≥ 18 years of age who presents with one of the following conditions:

  * Morphologically confirmed diagnosis of MDS with revised International Prognostic Scoring System (rIPSS) risk categories: intermediate, high and very high.
  * Morphologically confirmed diagnosis of CMML-2 with indication for azacitidine treatment.
  * CMML and MDS patient with response failure to HMA or therapy regimen including HMA.
  * Morphologically confirmed diagnosis of r/r AML following at least 1 line of prior therapies with indication for azacitidine treatment.
  * Morphologically confirmed diagnosis of AML in patients unfit for induction therapy with indication for azacitidine-venetoclax treatment.
* Leukocyte count < 20 x10^9/L (< 25 x10^9/L for newly diagnosed AML). Hydroxycarbamide use is permitted to meet this criterion in MDS and AML but not in CMML.
* Adequate renal function.
* Adequate liver function.

Exclusion Criteria:

* Patient with acute promyelocytic leukemia (APL) or myeloproliferative CMML as defined by leukocyte count > 13 x10^9/L.
* Eastern Cooperative Oncology Group (ECOG) performance status >2 (except newly diagnosed AML where ECOG 3 is allowed for patients < 75 years).
* Allogeneic transplantation less than 6 months prior screening.
* Patient with active auto-immune disorder (except type I diabetes, celiac disease, hypothyroidism requiring only hormone replacement, vitiligo, psoriasis, or alopecia).
* The patient requires systemic corticosteroid (≥10 mg/day prednisone or equivalent) or other immunosuppressive treatment.
* Less than 21 days since the last dose of intravenous anticancer chemotherapy or less than 14 days or five half-lives (whichever is shorter) from a small molecule targeted therapy or oral anticancer chemotherapy before the first study treatment.
* Any immunotherapy or investigational therapy within preceding 28 days from the first study treatment.
* Pregnant or lactating women.
* History of chronic ulcers or clinically relevant liver disease leading to Child Pugh Score C or higher.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 181 (Estimated)
Dates: Start 2022-06-02 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Reporting of incidence and frequency of dose limiting toxicities (DLTs). | From study start to end of Cycle 1 (each cycle is 28 days)
Frequency and severity based on NCI-CTCAE grading of treatment emergent AEs and serious adverse events (SAE). | From study start to 30 days after end of treatment (EOT)
Complete response (CR) rate for MDS and CMML-2. | From study start to 30 days after EOT
Overall response rate (ORR) for MDS and CMML failure to prior HMA. | From study start to 30 days after EOT
Complete remission with incomplete blood recovery (CRi) for r/r AML. | From study start to 30 days after EOT
Minimal residual disease (MRD) status for newly diagnosed AML. | From study start to 30 days after EOT

SECONDARY OUTCOMES:
Frequency and severity based on NCI-CTCAE grading of treatment emergent AEs and SAEs. | From study start to 30 days after EOT
Clinical efficacy measures based on progression free survival analyses defined as the time from study start to the date of documented disease progression or death from any cause, whichever occurs first, up to 2 years. | 24 months from study start
Clinical efficacy measures based on overall survival analyses defined as the length measured from study start to death from any cause up to 2 years. | 24 months from study start
Anti-bexmarilimab antibody positivity occurrence rate pre-dose and at defined timepoints during treatment. | 24 months from study start
Serum concentrations of bexmarilimab at defined timepoints pre-dose and post-dose of single and repeat bexmarilimab administrations using peripheral blood. | From study start to end of Cycle 2 (each cycle is 28 days)

CONTACTS AND LOCATIONS:
Overall Officials: Mika Kontro, MD, PhD, Principal Investigator — Helsinki University Central Hospital
Locations (10):
- United States (4):
  - City of Hope National Medical Center, Duarte, California
  - Yale Cancer Center, New Haven, Connecticut
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - University of Texas, MD Anderson Cancer Center, Houston, Texas
- Finland (4):
  - Helsinki University Hospital, Helsinki
  - Kuopio University Hospital, Kuopio
  - Oulu University Hospital, Oulu
  - Tampere University Hospital, Tampere
- United Kingdom (2):
  - The Christie NHS Foundation Trust, Manchester
  - Royal Cornwall Hospitals NHS Trust, Truro

REFERENCES:
- [Derived] Kontro M, Stein AS, Pyorala M, Rimpilainen J, Siitonen T, Ylitalo A, Fjallskog ML, Jalkanen J, Aakko S, Pawlitzky I, Hollmen M, Daver N. Bexmarilimab plus azacitidine for high-risk myelodysplastic syndrome and relapsed or refractory acute myeloid leukaemia: results from the dose-escalation part of a multicentre, single-arm, phase 1/2 trial. Lancet Haematol. 2025 Jul;12(7):e516-e528. doi: 10.1016/S2352-3026(25)00103-6. Epub 2025 May 28. PMID 40449509
- [Derived] Aakko S, Ylitalo A, Kuusanmaki H, Rannikko JH, Bjorkman M, Mandelin J, Heckman CA, Kontro M, Hollmen M. CLEVER-1 targeting antibody, bexmarilimab, supports HLA-DR expression and alters ex vivo responsiveness to azacitidine and venetoclax in myeloid malignancies. Sci Rep. 2025 May 14;15(1):16775. doi: 10.1038/s41598-025-01675-y. PMID 40369178